CLINICAL TRIAL: NCT03330262
Title: Head-Mounted Vibrotactile Prosthesis for Patients With Chronic Postural Instability
Acronym: BALCAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barron Associates, Inc. (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BALCAP1
Record Dates: First submitted 2017-05-11; First posted 2017-11-06 (Actual); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Vestibular Disorder; Dizziness
Keywords: Postural Instability; Balance Disorder; Balance Prosthesis; Dizziness
MeSH Terms: conditions — Vestibular Diseases; Dizziness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- BALCAP prosthesis, then Control (Experimental): Participants performed exercises daily at home wearing the BALCAP prosthesis for 6 weeks. After 6 weeks, participants performed the control condition (the same exercises without the BALCAP). Tests were performed before and after each 6-week period. Exercises included: (1) standing on a firm surface with feet apart, eyes open and closed; (2) standing on a firm surface with feet together, eyes open and closed; (3) standing on thick footing (e.g., multiple pairs of socks) with feet apart, eyes open and closed; (4) standing on thick footing with feet together, eyes open and closed; (5) standing in a modified Romberg position on a firm surface, eyes open and closed; (6) standing in a Romberg position on a firm surface, eyes open and closed; (7) walking on a firm surface eyes open; (8) walking with thick footing, eyes open; (9) walking with head turns and tilts, eyes open; and (10) walking around a room, with turns and movements other than straight forward walking, eyes open.
  Interventions: Device: BALCAP prosthesis
- Control, then BALCAP prosthesis (Experimental): Participants performed exercises daily at home for 6 weeks without wearing the BALCAP prosthesis (control), followed by another 6 weeks of the same exercises with the BALCAP prosthesis (intervention). Tests were performed before and after each 6 week period. Exercises included: (1) standing on a firm surface with feet apart, eyes open and closed; (2) standing on a firm surface with feet together, eyes open and closed; (3) standing on thick footing (e.g., multiple pairs of socks) with feet apart, eyes open and closed; (4) standing on thick footing with feet together, eyes open and closed; (5) standing in a modified Romberg position on a firm surface, eyes open and closed; (6) standing in a Romberg position on a firm surface, eyes open and closed; (7) walking on a firm surface eyes open; (8) walking with thick footing, eyes open; (9) walking with head turns and tilts, eyes open; and (10) walking around a room, with turns and movements other than straight forward walking, eyes open.
  Interventions: Device: BALCAP prosthesis

INTERVENTIONS:
Device: BALCAP prosthesis — The noninvasive BALCAP prosthesis offers uses six degrees-of-freedom (6-DOF) sensing to detect postural imbalance and actuate low-amplitude vibrotactile cues directly to the head to provide the wearer with feedback concerning head tilt in the pitch and roll plane.

SUMMARY:
The goal of this study is to evaluate a tactile prosthesis that provide individuals who have demonstrated chronic imbalance with help to maintain a correct sense of orientation with respect to the gravity and improve posture control.

DETAILED DESCRIPTION:
The goal of this study is to evaluate a tactile prosthesis that provide individuals who have demonstrated chronic imbalance with help to maintain a correct sense of orientation with respect to the gravity and improve posture control. Chronic imbalance leads to significant problems. This study is designed to evaluate a device which can potentially improve the balance of these patients.

The participant will be asked to come to Washington University on three occasions for approximately 2 hours. Between visits, they will be asked to use the device daily (intervention condition) or to not use the device (control condition) for a prescribed period of time doing different activities. They will be provided written instructions from a physical therapist that will be determined by their individual ability. The activities will be typical exercises that are given to people with balance disorders. After 6 weeks of home use, participants will return for the second visit, and will repeat the evaluation. They will then return home and complete the either the control or intervention condition (which was not done the first time) in a crossover design.

On their first visit (week 0; baseline) participants will be asked to complete the same kind of tests that evaluated the function of their balance system at the time of their diagnosis. They will have their eye movements recorded using goggles and an infra-red camera while the prosthesis is in place and providing vibration feedback. Computerized Dynamic Posturography (CDP) testing will require them to stand on a platform and perform tests (20 seconds each) with their eyes open or closed, with the platform moving or still, and/or with the visual surround either stable or moving. They will be fitted with a safety harness that will keep them from falling. Next the investigators will evaluate their ability to perform movement tasks while walking (walking down the hall, walking down the hall avoiding objects, changing speeds while walking, going up and down stairs etc). They will walk a 25-foot distance at a comfortable gait speed, and again at a maximum gait speed. Lastly, they will be asked to fill out questionnaires.

On their second and last visit, they will repeat the evaluations that were performed during the first visit.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory
* Chronic imbalance for at least 1 year
* Have reached a functional performance plateau with respect to balance performance
* Have a DGI score of <19
* Fall below age and gender matched normative data for gait speed

Exclusion Criteria:

* Subjects who are unwilling or unable to adhere to all study requirements, including completion of the training period, evaluation tests, and return to clinic for a follow-up visit.
* Women who are pregnant (women will self-report possible pregnancy).

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Parker, PHD, Principal Investigator — Barron Associates, Inc.
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BALCAP Prosthesis, Then Control: Participants were asked to perform a series of appropriate exercises daily at home wearing the BALCAP prosthesis for a period of 6 weeks. After the 6 weeks of the BALCAP intervention, participants performed the control condition (the same exercises without the BALCAP worn). Tests were performed before and after each 6 week period.
  The training exercises included: (1) standing on a firm surface with feet apart, eyes open and closed; (2) standing on a firm surface with feet together, eyes open and closed; (3) standing on thick footing (e.g., multiple pairs of socks) with feet apart, eyes open and closed; (4) standing on thick footing with feet together, eyes open and closed; (5) standing in a modified Romberg position on a firm surface, eyes open and closed; (6) standing in a Romberg position on a firm surface, eyes open and closed; (7) walking on a firm surface eyes open; (8) walking with thick footing, eyes open; (9) walking with head turns and tilts, eyes open; and (10) walking around a room, incorporating turns and movements other than straight forward walking, eyes open.
  BALCAP prosthesis: The noninvasive BALCAP prosthesis offers uses six degrees-of-freedom (6-DOF) sensing to detect postural imbalance and actuate low-amplitude vibrotactile cues directly to the head to provide the wearer with feedback concerning head tilt in the pitch and roll plane.
- Control, Then BALCAP Prosthesis: Participants were asked to perform a series of appropriate exercises daily at home for a period of 6 weeks without wearing the BALCAP prosthesis (control condition), followed by another 6 weeks of the same exercises with the BALCAP prosthesis (intervention condition). Tests were performed before and after each 6 week period.
  The training exercises included: (1) standing on a firm surface with feet apart, eyes open and closed; (2) standing on a firm surface with feet together, eyes open and closed; (3) standing on thick footing (e.g., multiple pairs of socks) with feet apart, eyes open and closed; (4) standing on thick footing with feet together, eyes open and closed; (5) standing in a modified Romberg position on a firm surface, eyes open and closed; (6) standing in a Romberg position on a firm surface, eyes open and closed; (7) walking on a firm surface eyes open; (8) walking with thick footing, eyes open; (9) walking with head turns and tilts, eyes open; and (10) walking around a room, incorporating turns and movements other than straight forward walking, eyes open.
Period: First Six Weeks
Arm/Group | BALCAP Prosthesis, Then Control | Control, Then BALCAP Prosthesis
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0
Period: Second Six Weeks
Arm/Group | BALCAP Prosthesis, Then Control | Control, Then BALCAP Prosthesis
Started | 7 | 6
Completed | 5 | 5
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BALCAP Prosthesis, Then Control | Control, Then BALCAP Prosthesis | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10.7) | 71.6 (11.5) | 69.7 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 6 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Difference in Dynamic Gait Index (DGI)
Description: This outcome compared the Dynamic Gait Index score when the BALCAP prosthesis was worn vs. when it was not worn at baseline in order to evaluate if there is an assistive benefit to wearing the device. The Dynamic Gait Index (DGI) is a clinical tool to assess gait, balance, and fall risk using various walking tasks. The range of scores is 0 to 24. A higher score is better. All participants performed this test at baseline both wearing the BALCAP and not wearing the BALCAP. This test does not measure a change in DGI score over time but compares the results of the test while wearing the BALCAP vs. not wearing the BALCAP during the same evaluation period (baseline).
Time Frame: Week 0 (baseline)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- All Participants: All participants performed the dynamic gait index at baseline both with and without the BALCAP prosthesis.
Arm/Group | All Participants
Number analyzed (Participants) | 13
units on a scale | 0.77 [0.16 to 1.38]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.018, Mixed Models Analysis

2. Secondary Outcome: Change in Computerized Dynamic Posturography: Equilibrium Score
Description: Change in Computerized Dynamic Posturography (CDP): equilibrium score. Computerized Dynamic Posturography is used to assess balance disorders using a balance platform. CDP is used to determine postural stability; it measures a patient's ability to maintain balance under multiple conditions by testing visual, vestibular, and somatosensory balance components of the body. The equilibrium score is an overall indicator of balance. A score of 100 represents perfect stability and a score of 0 indicates a loss of balance. A higher value is better. This test is intended to ascertain if there is a rehabilitative benefit of using the BALCAP instrument.
Time Frame: Before and after 6 weeks of either the intervention or the control condition
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- BALCAP Prosthesis: Participants who wore the BALCAP during exercises for either the first six weeks or the second six weeks of the protocol.
- Control: Participants who did not wear the BALCAP prosthesis when performing the exercises in either the first six weeks or the second six weeks of the protocol.
Arm/Group | BALCAP Prosthesis | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 5.94 [1.8 to 10.9] | 0.34 [-3.81 to 4.49]
Statistical Analysis 1: Comparison: BALCAP Prosthesis; Test type: Other — Ho: mean change = 0; p = 0.006, Mixed Models Analysis
Statistical Analysis 2: Comparison: Control; Test type: Other — Ho: mean change = 0; p = 0.869, Mixed Models Analysis

3. Secondary Outcome: Difference in Gait Speed
Description: The gait speed of each participant was measured over a 25-foot difference when wearing the BALCAP vs when not wearing the BALCAP. This test was performed on all participants at baseline prior to the home studies. A higher value represents faster gait speed. This test is intended to measure the assistive benefit of the BALCAP prosthesis.
Time Frame: Week 0 (baseline)
Measure: Mean (95% Confidence Interval); unit: meters/second
Groups:
- All Participants: All participants' 25-foot gait speed was measured while wearing the BALCAP prosthetic and while not wearing the BALCAP at baseline.
Arm/Group | All Participants
Number analyzed (Participants) | 13
meters/second | 0.03 [-0.05 to 0.11]
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.448, Mixed Models Analysis

4. Secondary Outcome: Change in Activities-specific Balance Confidence (ABC) Scale
Description: Change in Activities-specific Balance Confidence (ABC) Scale. The Activities-specific Balance Confidence Scale is a self-report questionnaire that measures an individual's confidence in performing activities without losing balance. The score range is from 0 to 100. A higher value is better.
Time Frame: Before and after 6 weeks of either the intervention or the control condition
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Control: Participants who did not wear the BALCAP during exercises for either the first six weeks or the second six weeks of the protocol.
Arm/Group | BALCAP Prosthesis | Control
Number analyzed (Participants) | 10 | 10
units on a scale | 6.04 [-5.45 to 17.53] | 1.39 [-10.10 to 12.88]
Statistical Analysis 1: Comparison: BALCAP Prosthesis; Test type: Other — This test evaluated whether the change in ABC was significant for the BALCAP condition##. Ho: mean = 0; p = 0.273, Mixed Models Analysis
Statistical Analysis 2: Comparison: Control; Test type: Other — This test evaluated if the change in ABC score was significant for the control group; p = 0.796, Mixed Models Analysis

5. Secondary Outcome: Change in Dizziness Handicap Inventory Score
Description: Change in Dizziness Handicap Inventory score. The Dizziness Handicap Inventory (DHI) is a common self-report quality of life measure for vestibular disorders. The score range is from 0 to 100 and a lower score is better. This test is intended to ascertain if there is a rehabilitative benefit of using the BALCAP instrument.
Time Frame: Before and after 6 weeks of either the intervention or the control condition
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BALCAP Prosthesis | Control
Number analyzed (Participants) | 10 | 10
units on a scale | -7.33 [-18.66 to 3.99] | 2.00 [-9.32 to 13.32]
Statistical Analysis 1: Comparison: BALCAP Prosthesis; Test type: Other — Ho: Mean change in score = 0; p = 0.189, Mixed Models Analysis
Statistical Analysis 2: Comparison: Control; Test type: Other — Ho: mean change = 0; p = 0.713, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: The 12 weeks of each participant's study.
Groups:
- BALCAP Prosthesis: Participants will be asked to perform a series of appropriate exercises daily at home wearing the BALCAP prosthesis for a period of 6 weeks. The training exercises will include: (1) standing on a firm surface with feet apart, eyes open and closed; (2) standing on a firm surface with feet together, eyes open and closed; (3) standing on thick footing (e.g., multiple pairs of socks) with feet apart, eyes open and closed; (4) standing on thick footing with feet together, eyes open and closed; (5) standing in a modified Romberg position on a firm surface, eyes open and closed; (6) standing in a Romberg position on a firm surface, eyes open and closed; (7) walking on a firm surface eyes open; (8) walking with thick footing, eyes open; (9) walking with head turns and tilts, eyes open; and (10) walking around a room, incorporating turns and movements other than straight forward walking, eyes open.
  BALCAP prosthesis: The noninvasive BALCAP prosthesis offers uses six degrees-of-freedom (6-DOF) sensing to detect postural imbalance and actuate low-amplitude vibrotactile cues directly to the head to provide the wearer with feedback concerning head tilt in the pitch and roll plane.
- Control: Participants will be asked to perform a series of appropriate exercises daily at home for a period of 6 weeks. The training exercises will include: (1) standing on a firm surface with feet apart, eyes open and closed; (2) standing on a firm surface with feet together, eyes open and closed; (3) standing on thick footing (e.g., multiple pairs of socks) with feet apart, eyes open and closed; (4) standing on thick footing with feet together, eyes open and closed; (5) standing in a modified Romberg position on a firm surface, eyes open and closed; (6) standing in a Romberg position on a firm surface, eyes open and closed; (7) walking on a firm surface eyes open; (8) walking with thick footing, eyes open; (9) walking with head turns and tilts, eyes open; and (10) walking around a room, incorporating turns and movements other than straight forward walking, eyes open.
Arm/Group | BALCAP Prosthesis | Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-25): https://cdn.clinicaltrials.gov/large-docs/62/NCT03330262/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT03330262/SAP_001.pdf